CLINICAL TRIAL: NCT01524302
Title: Pharmacodynamic of Ceftaroline and Levofloxacin Against Pathogens Associated With Community Acquired Bacterial Pneumonia (CABP)
Brief Title: Pharmacodynamic of Ceftaroline and Levofloxacin Against Pathogens Associated With Community Acquired Bacterial Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gary E. Stein, Pharm.D. (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Gary E. Stein, Pharm.D., Professor of Medicine and Pharmacology, Michigan State University
Organization: Michigan State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEF-MD-02
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Pneumonia, Bacterial; Community-acquired
Keywords: pneumonia; ceftaroline; community-aquired
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia | interventions — Ceftaroline; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levofloxacin (Active Comparator): Pharmacodynamics
  Interventions: Drug: Levofloxacin
- Ceftaroline (Active Comparator): Pharmacodynamics
  Interventions: Drug: Ceftaroline

INTERVENTIONS:
Drug: Ceftaroline — 600 mg Q12h
  Other Names: Teflaro
  Arms: Ceftaroline
Drug: Levofloxacin — 750 mg QD
  Other Names: Levaquin
  Arms: Levofloxacin

SUMMARY:
This study will further analyze the use of ceftaroline for CABP and compare its potential to eradicate bacterial pathogens to standard fluoroquinolone therapy. The enhanced spectrum of ceftaroline compared to levofloxacin may be further highlighted from this investigation.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant adults (≥ 18 years old) with suspected CABP admitted to the hospital for parenteral antibiotic therapy.
* All patients will have a creatinine clearance (CrCl) >50 ml/min.

Exclusion Criteria:

* pregnant or nursing patients,
* allergy to penicillin/cephalosporin antibiotics,
* allergy to fluoroquinolones,
* renal or hepatic failure, or have received an antimicrobial in past 96h.
* Patients who require antibiotics other than the study drugs will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Stein, Pharm.D., Principal Investigator — Michigan State University
Locations (1):
- Sparrow Hospital, Lansing, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levofloxacin | Ceftaroline
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin | Ceftaroline | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Full Range); unit: years] | 56 [26 to 72] | 52 [40 to 61] | 54 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Secondary Outcome: Mean (SD) Ceftaroline and Levofloxacin Pharmacokinetic Volume of Distribution Parameter in Community-Acquired Bacterial Pneumonia Patients
Description: To determine the serum pharmacokinetic volume of distribution of ceftaroline and levofloxacin in community-acquired bacterial pneumonia patients. We obtained blood at 2, 6 and 12 hours after at least 2 days of treatment and a 1-hr antibiotic infusion and measured these levels (mg/L)by LC/MS/MS assay.
Time Frame: 2, 6 and 12 hours after at least 2 days of treatment and a 1-hr antibiotic infusion
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Levofloxacin | Ceftaroline
Number analyzed (Participants) | 6 | 6
Liters | 92 (15) | 20.6 (5.2)

2. Secondary Outcome: Mean (SD) Doripenem Pharmacokinetic (PK) Clearance of Drug Parameter in Community-Acquired Bacterial Pneumonia Patients
Description: To determine the serum pharmacokinetic clearance of drug parameter of ceftaroline and levofloxacin in community-acquired bacterial pneumonia patients. We obtained blood at 2, 6 and 12 hours after at least 2 days of treatment and a 1-hr antibiotic infusion and measured these levels (mg/L)by LC/MS/MS assay.
Time Frame: 2, 6 and 12 hours after at least 2 days of treatment and a 1-hr antibiotic infusion
Measure: Mean (Standard Deviation); unit: liters per hour
Arm/Group | Levofloxacin | Ceftaroline
Number analyzed (Participants) | 6 | 6
liters per hour | 9.4 (3.1) | 7.3 (1.5)

3. Secondary Outcome: Mean (SD) Ceftaroline and Levofloxacin Pharmacokinetic (PK) Half Life Parameter in Community-Acquired Bacterial Pneumonia Patients
Description: To determine the serum pharmacokinetic half life parameter of ceftaroline and levofloxacin in community-acquired bacterial pneumonia patients. We obtained blood at 2, 6 and 12 hours after at least 2 days of treatment and a 1-hr antibiotic infusion and measured these levels (mg/L)by LC/MS/MS assay.
Time Frame: 2, 6 and 12 hours after at least 2 days of treatment and a 1-hr antibiotic infusion
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levofloxacin | Ceftaroline
Number analyzed (Participants) | 6 | 6
hours | 7.2 (1.4) | 1.9 (0.2)

4. Secondary Outcome: Mean (SD) Doripenem Pharmacokinetic (PK) Area Under Serum Curve (mg*h/L) Parameter in Community-Acquired Bacterial Pneumonia Patients.
Description: To determine the serum pharmacokinetic Area Under Serum Curve parameter of ceftaroline and levofloxacin in community-acquired bacterial pneumonia patients. We obtained blood at 2, 6 and 12 hours after at least 2 days of treatment and a 1-hr antibiotic infusion and measured these levels (mg/L)by LC/MS/MS assay.
Time Frame: 2, 6 and 12 hours after at least 2 days of treatment and a 1-hr antibiotic infusion
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Levofloxacin | Ceftaroline
Number analyzed (Participants) | 6 | 6
mg*hr/L | 87 (23) | 90 (15)

5. Primary Outcome: Serum Cidal Activity as Tested Against Staphylococcus Aureus Isolates and Reported as Ex-vivo Effect (Log Inhibition of Growth)
Description: Serum cidal activity of serum collected at 2 hour (levofloxacin) and 12 hour (ceftaroline) time points from the patients was tested against methyicillin-sensitive staphylococcus aureus isolates and the ex-vivo effect reported as log inhibition (logrithmic measurement of the decrease in microbiological growth).
  These staphylococcus aureus isolates had a range of minimum inhibitory concentrations (MIC) to Levofloxacin, 0.5, 1.0, 2.0, and 4.0 and the MIC's to Ceftaroline were 0.125, 0.19, 0.094, 0.094, respectively.
Time Frame: 2 hour (levofloxacin) and 12 hour (ceftaroline) after receiving the drug
Measure: Number; unit: Log inhibition
Groups:
- Log Inhibition of 0.5mg/L MIC Levofloxacin; Log Inhibition of 1.0mg/L MIC Levofloxacin; Log Inhibition of 2.0mg/L MIC Levofloxacin; Log Inhibition of 4.0mg/L MIC Levofloxacin: Measurement of the decrease in organism (Staphylococcus aureus) colony counts following exposure of serum containing Levofloxacin or Ceftaroline
Arm/Group | Log Inhibition of 0.5mg/L MIC Levofloxacin | Log Inhibition of 1.0mg/L MIC Levofloxacin | Log Inhibition of 2.0mg/L MIC Levofloxacin | Log Inhibition of 4.0mg/L MIC Levofloxacin
Number analyzed (Participants) | 12 | 12 | 12 | 12
Log inhibition
  Levofloxacin | 2 | 4 | 1 | 1
  Ceftaroline | 3 | 5 | 3 | 3

ADVERSE EVENTS:
Arm/Group | Levofloxacin | Ceftaroline
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No